CLINICAL TRIAL: NCT06324786
Title: Brain Mechanisms of Reducing Polysubstance Use Following a Novel Body-mind Intervention 2
Brief Title: Brain Mechanisms of Reducing Polysubstance Use
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2024 IBMT NF
Record Dates: First submitted 2024-03-06; First posted 2024-03-22 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Multiple Drug Use

STUDY DESIGN:
Intervention Model Description: mindfulness or/and active/sham neurofeedback
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IBMT (Experimental): An evidence-based preventive intervention - integrative body-mind training (IBMT) has shown positive effects in reducing stress and improving self-control and brain plasticity. It has bodifulness and mindfulness components.
  Interventions: Behavioral: IBMT
- NF (Experimental): An evidence-based intervention - NF can not only provide real-time feedback for practice but also target the self-control networks, suggesting the possibility of augmenting IBMT effects via NF.
  Interventions: Behavioral: NF
- IBMT + NF (Experimental): The combined IBMT and NF also show positive effects in reducing substance use.
  Interventions: Behavioral: IBMT; Behavioral: NF
- Sham NF (Sham Comparator): Sham NF has the same settings as the active NF but does not have correct parameters of stimulation.
  Interventions: Behavioral: NF

INTERVENTIONS:
Behavioral: IBMT — IBMT is an effortless mindfulness technique
  Arms: IBMT; IBMT + NF
Behavioral: NF — NF is a mental training technique.
  Arms: IBMT + NF; NF; Sham NF

SUMMARY:
The proposed study will test whether neurofeedback (NF) could optimize integrative body-mind training (IBMT) practice.

DETAILED DESCRIPTION:
The proposed study will test whether real-time NF could optimize IBMT practice and improve effects in reducing polysubstance use through targeting self-control networks in the brain.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Free of any psychiatric diagnoses or medication (besides a substance use disorder (SUD) to alcohol, tobacco, or cannabis)
* In the past month, at least 4 episodes of heavy episodic drinking; at least 3 occasions of cannabis use; and daily cigarette use for at least the past month
* Normal or corrected-to-normal vision
* Written informed consent
* No previous meditation or NF experiences

Exclusion Criteria:

* Any psychiatric diagnoses other than an SUD
* Medical disorder(s) that may affect the central nervous system; medications that affect the central and autonomic nervous system; or a positive pregnancy test result (females)
* Excluding cannabis, evidence of recent (past month) illicit drug use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Intervention effects on brain function using Functional Magnetic Resonance Imaging (fMRI) | The outcome measures are assessed in-person at baseline, 2-4 weeks and 3 months
  Brain connectivity changes such as anterior and posterior cingulate cortex measured by fMRI resting state imaging
Intervention effects on brain white matter using fMRI | The outcome measures are assessed in-person at baseline, 2-4 weeks and 3 months
  Brain white matter changes such as anterior and posterior cingulate cortex measured by fMRI diffusion tensor imaging
Intervention effects on brain grey matter using fMRI | The outcome measures are assessed in-person at baseline, 2-4 weeks and 3 months
  Brain volume changes such as anterior and posterior cingulate cortex measured by fMRI structural imaging

SECONDARY OUTCOMES:
Intervention effects on addiction behavior using substance use questionnaires in PhenX Toolkit | The outcome measures are assessed in-person at baseline, 2-4 weeks and 3 months
  Intervention leads to a significant reduction in craving and substance use measured by substance use questionnaires in PhenX Toolkit

CONTACTS AND LOCATIONS:
Locations (1):
- YiYuan Tang, Phoenix, Arizona, United States